CLINICAL TRIAL: NCT00762684
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel Study of the Safety and Efficacy of TAK-559 Compared to Placebo in the Treatment of Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety Study of TAK-559 in Treating Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Hepatic safety signal identified.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-04-TL-559-028; U1111-1127-7965 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — (E)-4-(4-((5-methyl-2-phenyl-1,3-oxazol-4-yl)methoxy)benzyloxyimino)-4-phenylbutyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-559 32 mg QD (Experimental)
  Interventions: Drug: TAK-559
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-559 — TAK-559 32 mg, tablets, orally, once daily for up to 26 weeks.
  Arms: TAK-559 32 mg QD
Drug: Placebo — TAK-559 placebo-matching tablets, orally, once daily for up to 26 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study was to determine the safety and efficacy of TAK-559, once daily (QD), in treating subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Insulin is a primary regulator of blood glucose concentrations. A subnormal response to circulating insulin levels at target tissues leads to a decrease in insulin-mediated glucose uptake. Insulin resistance is associated with normal to high insulin levels and is often accompanied by dyslipidemia, a disruption in lipid metabolism resulting in increased triglycerides and low-density lipoprotein levels as well as decreased high-density lipoprotein levels in patients with type 2 diabetes mellitus. In the early stages of insulin resistance, a compensatory mechanism of increased insulin secretion by the pancreas maintains normal to near-normal glucose levels. Once the pancreas fails to maintain the increased insulin output, overt type 2 diabetes mellitus occurs.

TAK-559 is a novel oxyiminoalkanoic acid under investigation for use as an oral agent in the treatment of patients with type 2 diabetes mellitus. TAK-559 has partial peroxisome proliferator-activated receptor-alpha agonist activity, potent peroxisome proliferator-activated receptor-alpha activity, and modest peroxisome proliferator-activated receptor-gamma activity at high concentrations in nonclinical models.

This study was designed to evaluate the safety and glycemic control of TAK-559 in patients with type 2 diabetes mellitus whose symptoms were managed by diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Was diagnosed with type 2 diabetes mellitus using American Diabetes Association diagnostic criteria, and on a stable dose of an oral anti-diabetic monotherapy prior to Screening A.
* Had a glycosylated hemoglobin level greater than or equal to 8.0% and less than or equal to 10.0% at Screening B.
* Had a fasting plasma glucose greater than or equal to 126 mg/dL (7.0 mmol/L) at Screening B.
* Was taking a stable dose of at least 10 mg of glyburide for at least 10 days prior to Screening B.
* Had a stable or worsening self-monitoring blood glucose level while taking glyburide.
* Had a low-density lipoprotein less than 160 mg/dL (4.1 mmol/L) at Screening A.
* Had a body mass index less than or equal to 45 kg/m2 at Screening A.
* Was willing to be counseled by the investigator or designee to follow an individualized, weight-maintaining diet during the study period.
* Had evidence of insulin secretory capacity as demonstrated by a C-peptide concentration of greater than or equal to 1.5 ng/mL (0.50 nmol/L) at Screening A, and if necessary, after a repeat at Screening B.
* Was able to perform daily self-monitoring blood glucose tests throughout the study.
* Had a normal thyroid-stimulating hormone level of less than 5.5 uIU/mL (5.5 mIU/L) and greater than or equal to 0.35 uIU/mL (0.35 mIU/L) at Screening A.
* Was in good health as determined by a physician (ie, via medical history and physical examination), other than a diagnosis of type 2 diabetes mellitus.
* Had fasting clinical laboratory evaluations within the normal reference range for the testing laboratory, or if not, the results must be deemed not clinically significant by the investigator prior to Randomization.
* Females were post menopausal, surgically sterile, or using adequate contraception.

Exclusion Criteria:

* Had been diagnosed with type 1 diabetes mellitus, hemochromatosis, or has a history of ketoacidosis.
* Had any condition known to invalidate glycosylated hemoglobin results (eg, hemolytic states, hemoglobinopathies).
* Was required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Insulin
  * Oral anti-diabetics other than TAK-559 (including sulfonylureas other than glyburide, alpha-glucosidase inhibitors, metformin)
  * Systemic corticosteroids
  * Warfarin
  * Rifampin
  * St. John's Wort.
  * Thiazolidinediones
  * Peroxisome proliferator-activated receptor agonists
  * Nicotinic Acid
  * Fibrates
* Had a history of myocardial infarction, coronary angioplasty or bypass graft, unstable angina pectoris, transient ischemic attacks, clinically significant abnormal electrocardiogram, or documented cerebrovascular accident within 6 months prior to Screening A.
* Had abdominal, thoracic, or vascular surgery within 6 months prior to Screening A that in the investigator's opinion would warrant exclusion from the study.
* Had a creatine phosphokinase value greater than 3 times the upper limit of normal at Screening A. The creatine phosphokinase value can be retested prior to Randomization if elevated.
* Had persistent unexplained microscopic or macroscopic hematuria or a history of bladder cancer.
* Had a triglyceride level greater than 500 mg/dL (5.6 mmol/L) at Screening A.
* Had any alteration in allowed lipid lowering medication (dose or drug) within 2 months of Randomization, if applicable.
* Had donated and/or received any blood or blood products within 3 months prior to Randomization.
* Had a history of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within 2 years prior to Randomization.
* Had a systolic BP greater than 140 mm Hg or a diastolic blood pressure of greater than 95 mm Hg at Screening B.
* Had significant cardiovascular disease including but not limited to, New York Heart Association Functional (Cardiac) Classification III or IV.
* Had a previous history of cancer, other than basal cell or stage 1 squamous cell carcinoma of the skin, that has not been in remission within 5 years prior to Randomization.
* Had an alanine transaminase or aspartate transaminase level greater than 3 times the upper limit of normal, active liver disease, or jaundice at Screening A.
* Had a positive human immunodeficiency virus, hepatitis B surface antigen, or hepatitis B e antigen test at Screening A.
* Had any other serious disease or condition at Screening A or at Randomization that might affect life expectancy or make it difficult to successfully manage and follow the patient according to the protocol.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-11; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycosylated hemoglobin. | Final Visit.

SECONDARY OUTCOMES:
Change from baseline in glycosylated hemoglobin. | Weeks 4, 8, 12, 16 and 20
Change from baseline in fasting plasma glucose. | Weeks 2, 4, 8, 12, 16, 20 and Final Visit
Change from baseline in serum insulin. | Weeks 4, 12, 16, 20 and Final Visit.
Change from baseline in C-peptide. | Weeks 4, 12, 16, 20 and Final Visit.
Change from baseline in triglycerides. | Weeks 12, 16, 20 and Final Visit.
Change from baseline in total cholesterol. | Weeks 12, 16, 20 and Final Visit.
Change from baseline in high-density lipoprotein. | Weeks 12, 16, 20 and Final Visit.
Change from baseline in low-density lipoprotein. | Weeks 12, 16, 20 and Final Visit.
Change from baseline in very-low-density lipoprotein. | Weeks 12, 16, 20 and Final Visit.
Change from base line in apolipoproteins A1 and B 100. | Final Visit
Change from baseline in free fatty acids. | Weeks 12, 16, 20 and Final Visit.
Change from baseline in thrombosis marker (plasminogen activator inhibitor-1) | Weeks 4, 12, 16, 20 and Final Visit
Change from baseline in thrombosis marker (fibrinogen) | Weeks 4, 12, 16, 20 and Final Visit
Change from baseline in inflammation marker (Interleukin-6). | Weeks 4, 12, 16, 20 and Final Visit
Change from baseline in inflammation marker (C-reactive protein). | Weeks 4, 12, 16, 20, and Final Visit
Change from baseline in urinary albumin to creatinine ratio. | Weeks 12, 16, 20 and Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda